CLINICAL TRIAL: NCT01575145
Title: Helping Hospitalized Patients Quit Smoking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David Warner, Associate Director of Clinical and Translational Research, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-002207
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Tobacco Abuse Cigarette

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quitline facilitation intervention (Experimental): brief quitline facilitation intervention given
  Interventions: Behavioral: Quitline facilitation intervention
- Stop-smoking intervention (Active Comparator): brief review of tips to maintain smoking abstinence, using brochure
  Interventions: Behavioral: Brief stop-smoking intervention

INTERVENTIONS:
Behavioral: Quitline facilitation intervention — brief quitline facilitation intervention
  Arms: Quitline facilitation intervention
Behavioral: Brief stop-smoking intervention — brief review of tips to help maintain smoking abstinence, using brochure
  Arms: Stop-smoking intervention

SUMMARY:
The study is being done to determine whether an in-hospital intervention using a brief intervention to facilitate quitline utilization will increase quitline utilization by hospitalized smokers, and will increase post hospital discharge smoking abstinence rates.

Study participants will be randomized to receive either a brief quitline facilitation intervention , or a control intervention of a brief stop-smoking message.

The study will also compare healthcare costs and utilization in the first six months following hospitalization between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Current smoker, Resident of Olmsted County, Inpatient admission to St. Marys or Rochester Methodist Hospital, Able to participate fully in all study aspects, Available for follow-up

Exclusion Criteria:

Current active treatment for tobacco use initiated prior to hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence tobacco abstinence at 6 months after hospitalization | 6 months after hospitalization

SECONDARY OUTCOMES:
Self-efficacy | Immediately after the delivery of the brief intervention (day of enrollment)
  Use of Smoking Self-Efficacy Questionnaire 12

CONTACTS AND LOCATIONS:
Overall Officials: David Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Nolan MB, Borah BJ, Moriarty JP, Warner DO. Association between smoking cessation and post-hospitalization healthcare costs: a matched cohort analysis. BMC Health Serv Res. 2019 Dec 2;19(1):924. doi: 10.1186/s12913-019-4777-7. PMID 31791307
- [Derived] Nolan MB, Borah BJ, Moriarty JP, Warner DO. Economic Analysis of a Geographically Defined Cohort of Hospitalized Patients Who Smoke. Mayo Clin Proc. 2018 Aug;93(8):1034-1042. doi: 10.1016/j.mayocp.2018.02.022. Epub 2018 Jul 4. PMID 30078410